CLINICAL TRIAL: NCT04014322
Title: The Effect of Electronic Cigarette Use on Smoking Behaviors and Smoking-related Factors Among Smokers Receiving Outpatient Psychiatric Treatment
Brief Title: The Effect of Electronic Cigarette Use on Smoking Behaviors Among Smokers Receiving Outpatient Psychiatric Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fordham University (Other)
Collaborators: Montefiore Medical Center (Other); Dartmouth College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1089
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Smoking; Psychiatric Disorders
Keywords: electronic cigarette use; smoking behavior
MeSH Terms: conditions — Tobacco Smoking; Mental Disorders; Vaping; Smoking | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- E-cigarette (Experimental): All participants will be instructed to switch completely from combustible cigarettes to e-cigarettes for the next 8weeks. They will be assessed at baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks.
  Interventions: Other: E-cigarette

INTERVENTIONS:
Other: E-cigarette — All participants will be provided with 8 weeks of e-cigarettes at no cost based on self-report of regular cigarette use.
  All participants will receive a total of 8-10 remote counseling sessions (via phone or video conference) and during which they will discuss ways to switch from smoking cigarettes to exclusively using e-cigarettes, barriers and strategies to overcome them. (All participants will receive sessions at baseline, 2 days, 7 days, 2 weeks, 3 weeks, and 4 weeks, 6 weeks , and 8 weeks after the baseline assessment. Two additional sessions at 5 weeks and 7 weeks (after the baseline assessment) will be provided to those who are still smoking combustible cigarettes at 4-week assessment.)

SUMMARY:
This study aims to establish the feasibility and acceptability of a project designed to investigate the impact of electronic cigarette use on combustible cigarette smoking and smoking-related factors among smokers with psychiatric disorders, a high-risk population, who are not yet ready to quit smoking. All participants will be instructed to switch completely from combustible cigarettes to e-cigarettes for the next 8 weeks. They will be assessed at baseline, 2 weeks, 4 weeks, 8 weeks and 12 weeks.

DETAILED DESCRIPTION:
In recent years, the prevalence of e-cigarette use has rapidly increased, especially among those with psychiatric conditions, and the risks and potential benefits of e-cigarette use have been the topic of much debate. More research is needed to understand the impact of e-cigarette use on smoking behavior and smoking-related cognitions among individuals with psychiatric conditions.

This study will investigate the effects of e-cigarette use on cigarette smoking and motivation/readiness to quit among smokers with psychiatric disorders who are not yet ready to quit smoking. A total of 50 adult daily cigarette smokers who are receiving outpatient psychiatric treatment and not yet ready to quit smoking will be recruited. All participants will be instructed to switch completely from combustible cigarettes to e-cigarettes for the next 8 weeks. E-cigarettes will be provided to participants at no cost. Participants will also be asked to complete 5 (remote and in-person) assessment sessions (i.e., baseline, 2-week, 4-week, 8-week and 12-week follow-ups).

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* English-speaking,
* current daily smokers (i.e., at least 5 cigarettes/day)
* have been daily smokers at least for 6 months
* attended a minimum of 2 treatment visits in the past 12 months at Montefiore Behavioral Health Center
* have at least one psychiatric disorder (other than substance use disorders),
* willing to try switching to use e-cigarettes (provided by the research team) exclusively for a total of 8 weeks,
* those who are not yet ready to quit smoking,
* for women of childbearing age, willingness to use contraception during the study.

Exclusion Criteria:

* acute psychiatric symptomatology which precludes study participation including current active suicidal ideation
* current diagnosis of dementia or cognitive impairment sufficient to impair provision of informed consent or study participation
* patient's inability to provide consent for study participation due to his/her inability to demonstrate an understanding of study procedures as contained in the statement of informed consent, after no more than two explanations
* current clinical diagnosis of intellectual development disorder
* current regular use of other tobacco products or combustible marijuana
* current (non-nicotine) substance use disorder and current substance use (in the past month)
* current effort to quit smoking or current use of pharmacotherapy (in the past month) to quit smoking,
* pregnant, breastfeeding, or planning to become pregnant within 6 months, current unstable cardiovascular disease,
* current unstable pulmonary disease (i.e., an ER visit or hospitalization due to pulmonary issues in the past 6 month or current use of oxygen therapy),
* patient does not have a stable home address where the research team could reliably reach patient
* household members are currently participating or have participated in this research study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the number of combustible cigarettes smoked per day | Baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks
  The average number of cigarettes smoked per day
Changes in Carbon Monoxide Level | Baseline,2 weeks, 4 weeks, 8 weeks, 12 weeks
  Changes in Carbon monoxide level measured with a breath carbon monoxide monitor
Changes in Nicotine Dependence | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Fagerstrom Test of Cigarette Dependence
Changes in the use of e-cigarettes | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Changes in the use of e-cigarettes
Rates of those who completely switched to e-cigarettes | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Rates of those who completely switched to e-cigarettes

SECONDARY OUTCOMES:
Changes in Motivation/Readiness to Quit Smoking | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Thoughts about Abstinence Scale & Contemplation Ladder
Changes in Withdrawal Symptoms | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Minnesota Nicotine Withdrawal Scale

CONTACTS AND LOCATIONS:
Overall Officials: Haruka Minami, Ph.D., Principal Investigator — Fordham University
Locations (1):
- Montefiore Behavioral Health Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No